CLINICAL TRIAL: NCT03379012
Title: Phase 2 Randomized Study of Efficacy and Safety of Testosterone in Metastatic Renal Cell Carcinoma Patients With Fatigue
Brief Title: Testosterone in Metastatic Renal Cell Carcinoma Patients
Acronym: FARETES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCRB08022016
Record Dates: First submitted 2017-10-13; First posted 2017-12-20 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — testosterone undecanoate; Sunitinib; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (2):
- Testosterone and Targeted therapy (Experimental): Testosterone undecanoate (Nebido®) and Targeted therapy (sunitinib or pazopanib)
  Interventions: Drug: Testosterone undecanoate and sunitinib or pazopanib
- Control (Active Comparator): Targeted therapy (sunitinib or pazopanib) only
  Interventions: Drug: Testosterone undecanoate and sunitinib or pazopanib

INTERVENTIONS:
Drug: Testosterone undecanoate and sunitinib or pazopanib — Testosterone undecanoate (Nebido®) 1,000 mg (4 ml) intramuscular deeply, once before targeted therapy (sunitinib 50 mg 4/2 or pazopanib 800 mg daily)

SUMMARY:
Purpose

To determine efficacy and safety of Testosterone in male patients with metastatic renal cell carcinoma and fatigue receiving targeted therapy or checkpoint inhibitors.

DETAILED DESCRIPTION:
Fatigue is a frequent symptom of metastatic renal cell carcinoma (RCC), and most common adverse event of targeted and immunotherapy.

In Phase 3 pivotal studies, 56% (9%, grade 3-4), 54% (11%, grade 3), 37% (10%, grade 3-4) and 20% (2%, grade 3) of patients had fatigue during the therapy of cabozantinib, sunitinib, axitinib or pazopanib, respectively. 59% (14%, grade 3) and 31% (5%, grade 3) of patients treated with lenvatinib/everolimus and everolimus had fatigue in registrational trials. Finally, 33% (2%, grade 3-4) of patients that received nivolumab had fatigue in CheckMate 025 study.

Testosterone may help to relieve fatigue associated with the use of tyrosine kinase, mTOR or checkpoint inhibitors. Additionally, testosterone could impact on poor prognostic factors of RCC (anemia, ECOG performance status, serum calcium). This will be first clinical trial which evaluates safety and efficacy of Testosterone in RCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven clear cell renal cell carcinoma;
2. CT-confirmed metastatic measurable disease;
3. First-line sunitinib or pazopanib treatment with fatigue;
4. Low level of testosterone;

4. Male, 18 years and older; 5. Normal PSA level

Exclusion Criteria:

1. Prostate and other cancers history
2. Hypothyroidism
3. History of serious cardiac arrhythmia, congestive heart failure, angina pectoris, or other severe cardiovascular disease (i.e., New York Heart Association class III or IV)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 60 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Fatigue | 3 months
  Difference in mean change of Fatigue from baseline score with testosterone vs. without testosterone.

SECONDARY OUTCOMES:
Safety and tolerability | 3 months
  Safety and tolerability of testosterone (CTCAE v.4.03)
Quality of life | 3 months
  Health-related quality of life (NCCN-FACT FKSI-19 (Version 2)
Overall rate of adverse events | 3 months
  Overall rate of adverse events related with TKI treatment (CTCAE v.4.03)
Testosterone serum concentrations | 12 weeks
  Maximum and minimum total testosterone serum concentrations following dose administration at week 12
Red blood cell count and Hemoglobin concentration | 12 weeks
  Change in Red blood cell count and Hemoglobin concentration following dose administration at week 12
Serum calcium concentration | 12 weeks
  Change in serum calcium concentration following dose administration at week 12
ECOG PS | 3 months
  ECOG Performance status
Overall survival | 2 years
  Time from randomization to death

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - A.I. Kryzhanovsky Krasnoyarsk Cancer Center, Krasnoyarsk
  - Kidney Cancer Research Bureau, Moscow
  - RUDN University, Moscow
  - City Clinical Oncology Center, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- [Background] Motzer RJ, Escudier B, Tomczak P, Hutson TE, Michaelson MD, Negrier S, Oudard S, Gore ME, Tarazi J, Hariharan S, Chen C, Rosbrook B, Kim S, Rini BI. Axitinib versus sorafenib as second-line treatment for advanced renal cell carcinoma: overall survival analysis and updated results from a randomised phase 3 trial. Lancet Oncol. 2013 May;14(6):552-62. doi: 10.1016/S1470-2045(13)70093-7. Epub 2013 Apr 16. PMID 23598172
- [Background] Sternberg CN, Hawkins RE, Wagstaff J, Salman P, Mardiak J, Barrios CH, Zarba JJ, Gladkov OA, Lee E, Szczylik C, McCann L, Rubin SD, Chen M, Davis ID. A randomised, double-blind phase III study of pazopanib in patients with advanced and/or metastatic renal cell carcinoma: final overall survival results and safety update. Eur J Cancer. 2013 Apr;49(6):1287-96. doi: 10.1016/j.ejca.2012.12.010. Epub 2013 Jan 12. PMID 23321547
- [Background] Motzer RJ, Hutson TE, Glen H, Michaelson MD, Molina A, Eisen T, Jassem J, Zolnierek J, Maroto JP, Mellado B, Melichar B, Tomasek J, Kremer A, Kim HJ, Wood K, Dutcus C, Larkin J. Lenvatinib, everolimus, and the combination in patients with metastatic renal cell carcinoma: a randomised, phase 2, open-label, multicentre trial. Lancet Oncol. 2015 Nov;16(15):1473-1482. doi: 10.1016/S1470-2045(15)00290-9. Epub 2015 Oct 22. PMID 26482279
- [Background] Motzer RJ, Escudier B, Oudard S, Hutson TE, Porta C, Bracarda S, Grunwald V, Thompson JA, Figlin RA, Hollaender N, Kay A, Ravaud A; RECORD-1 Study Group. Phase 3 trial of everolimus for metastatic renal cell carcinoma : final results and analysis of prognostic factors. Cancer. 2010 Sep 15;116(18):4256-65. doi: 10.1002/cncr.25219. PMID 20549832
- [Background] Tomita Y, Fukasawa S, Shinohara N, Kitamura H, Oya M, Eto M, Tanabe K, Kimura G, Yonese J, Yao M, Motzer RJ, Uemura H, McHenry MB, Berghorn E, Ozono S. Nivolumab versus everolimus in advanced renal cell carcinoma: Japanese subgroup analysis from the CheckMate 025 study. Jpn J Clin Oncol. 2017 Jul 1;47(7):639-646. doi: 10.1093/jjco/hyx049. PMID 28419248